CLINICAL TRIAL: NCT03176355
Title: Evaluation of Intraoperative Mitomycin C in Surgical Management of Lacrimal Sac Mucocele
Brief Title: Intraoperative Mitomycin C in Lacrimal Sac Mucocele
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Farag Khalil Ibrahiem, Lecturer of ophthalmology, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Minia Hospital
Record Dates: First submitted 2017-05-28; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Lacrimal Mucocele

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic dacryocystitis patients (Other)
  Interventions: Procedure: Canaliculo- Dacryocystorhinostomy

INTERVENTIONS:
Procedure: Canaliculo- Dacryocystorhinostomy — Bypass lacrimal passage obstruction by opening a shunt between the lacrimal sac and the nasal mucosa

SUMMARY:
30 patients had lacrimal sac mucocele and dacryocystorhinostomy was done for them with intraoperative mitomycin C was added to decrease postoperative fibrosis and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Lacrimal sac mucocele

Exclusion Criteria:

* Paediatric patients (less than 16 years old).
* Previous lacrimal passage procedure.
* Neoplasms as secondary causes of obstruction.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03-23 (Actual); Primary Completion 2012-01-07 (Actual); Study Completion 2013-01-07 (Actual)

PRIMARY OUTCOMES:
Disappearance of the watering of the eye reported by the patients and by fluorescein disappearance test | 1 month
  Patency of the lacrimal passage
Disappearance of lacrimal sac swelling | 1 month
  No evident swelling in the medial side of the eye